CLINICAL TRIAL: NCT00456300
Title: The Role of Exenatide in Type 1 Diabetes Mellitus
Brief Title: Role of Exenatide in Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Rubina Heptulla, Principal Investigator, Montefiore Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H-16488
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Type 1 Diabetes
Keywords: Hypoglycemia; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia; Hyperglycemia | interventions — Exenatide; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Exenatide 1.25 mcg + Insulin (Experimental): In each intervention arm the participant receives a different dose of Exenatide along with Insulin as a single subcutaneous injection
  Interventions: Drug: Exenatide; Drug: Insulin
- Exenatide 2.5 mcg + Insulin (Experimental): In each intervention arm the participant receives a different dose of Exenatide along with Insulin as a single subcutaneous injection
  Interventions: Drug: Exenatide; Drug: Insulin
- Insulin (Active Comparator): Each subject received a baseline study with insulin alone
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Exenatide — In each intervention arm the participant receives a different dose (1.25 or 2.5 mcg) of exenatide.
  Other Names: Byetta
  Arms: Exenatide 1.25 mcg + Insulin; Exenatide 2.5 mcg + Insulin
Drug: Insulin — Each subject received a baseline study with insulin alone

SUMMARY:
The purpose of this study is to see if giving exenatide and insulin before a meal would lower blood sugars after the meal. This study may help in developing new treatments to help control high blood sugars after meals. This may help improve overall blood sugar control and prevent the long-term effects of diabetes.

DETAILED DESCRIPTION:
A large study in people with type 1 diabetes (T1DM) showed that lowering blood sugars stopped or delayed the occurrence of health problems. As a result of the study, treatment should try to control blood sugars as near to normal as safely possible.

In people without diabetes, the "after meal" blood sugar level is very carefully controlled. Insulin (the hormone that lowers blood sugar) and glucagon (hormone that raises blood sugar) play a key role in keeping this careful balance. It is now known that a substance made by the body called GLP-1 also helps with this careful balance. Glucagon like peptide-1 works in four ways. First, it helps to stimulate the cells in the pancreas to produce more insulin. Secondly, it helps to "dampen" the glucagon response (glucagon is released after a meal and causes the blood sugar to rise). Thirdly, Glucagon like peptide-1 delays the digestion of food in the stomach. Lastly, it seems to "dampen" the appetite, which causes a person to eat less.

Exenatide is a medication that works very similar to Glucagon like peptide-1. Exenatide is FDA approved for use in adults.

Study Design: Followed by a baseline study with insulin alone, subjects were randomized to two different doses of exenatide (1.25 and 2.5 µ,g), administered in a double-blinded randomized controlled manner, along with insulin as a single subcutaneous injection. Studies were at least 3 weeks apart.

Baseline: At 0800 h, the pre-breakfast insulin bolus was administered based on patient's usual insulin-to-carbohydrate ratio. Post-bolus, subjects drank 12 ounces of a standard liquid meal (Boost High Protein Drink, 360 calories, 50 g carbohydrates, and 12 g fat), enriched with 1 g of [13C] glucose within 10 min. Breath samples for 13CO2 analysis were collected in duplicates at 17 time points until 1300 h. Usual insulin basal rates or glargine were maintained during study.

On the days subjects received the study drug of 1.25 µ,g (~0.02 µ,g/kg) or 2.5 µ,g (~0.04 µ,g/kg) exenatide along with insulin, the prandial insulin was reduced by 20%.

Measurements: Plasma glucose was measured using a bedside YSI glucose analyzer (2300 Stat Plus; Yellow Springs Instruments, Yellow Springs, OH) throughout the study at regularly timed intervals. Delta plasma glucose area under the curve (AUC0 -120) was measured for the exenatide treated groups vs. insulin monotherapy.

ELIGIBILITY:
Inclusion Criteria:

***Subjects must be patients of the Texas Children's Hospital Diabetes Care Center***.

All of the following criteria must be met:

1. Between 12-21 years of age at the time of enrollment.
2. Have been diagnosed with Type 1 diabetes for at least 1 year and in good control (HbA1C less than 8.5%).
3. Subjects must be otherwise healthy except for the Type 1 Diabetes and treated hypothyroidism.
4. Menstruating women must have a negative pregnancy test.
5. Hemoglobin equal to or greater than 12 g/dL before each study.
6. Weight greater than 44 kg.
7. Tanner stage greater than 3

Exclusion Criteria:

1. Any chronic disease: leukemia, asthma, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis etc or on treatment that might directly or indirectly affect glucose homeostasis, except for diabetes and hypothyroidism; stable on medications.
2. Lack of a supportive family environment as detected by the clinicians and/or social workers.
3. Positive pregnancy test in menstruating young women.
4. BMI greater than 90th percentile for age or less than 10th percentile for age.
5. Lactating and nursing mothers.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubina Heptulla, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Texas Children's Hospital/ Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raman VS, Mason KJ, Rodriguez LM, Hassan K, Yu X, Bomgaars L, Heptulla RA. The role of adjunctive exenatide therapy in pediatric type 1 diabetes. Diabetes Care. 2010 Jun;33(6):1294-6. doi: 10.2337/dc09-1959. Epub 2010 Mar 23. PMID 20332358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 subjects were enrolled into the study. Of these, 9 subjects were randomized and only 8 subjects completed this three part study. These subjects were recruited from the diabetes clinics.
Pre-assignment Details: Two subjects failed screening and could not be randomized to particiapate.
Groups:
- Insulin First, Then Exenatide1.25 mcg, Then Exenatide 2.5 mcg: Each of the eight study subjects underwent three study visits at-least 3 weeks apart; at each visit receiving either Insulin alone, Exenatide 1.25 mcg + Insulin or Exenatide 2.5 mcg + Insulin
- Insulin First, Then Exenatide 2.5 mcg, Then Exenatide 1.25 mcg: Each of the eight study subjects underwent three study visits at-least 3 weeks apart; at each visit receiving either Insulin alone, Exenatide 2.5 mcg + Insulin or Exenatide 1.25 mcg + Insulin
Period: Overall Study
Arm/Group | Insulin First, Then Exenatide1.25 mcg, Then Exenatide 2.5 mcg | Insulin First, Then Exenatide 2.5 mcg, Then Exenatide 1.25 mcg
Started ("Started" means recruited, not enrolled.) | 5 | 4
Completed | 4 | 4
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Following the baseline study with insulin, Participants were randomized to receive either Exenatide 1.25 mcg or Exenatide 2.5 mcg
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Plasma Glucose Area Under the Curve (AUC) for Blood Glucose Concentration in the Exenatide 1.25 mcg or Exenatide 2.5 mcg Treated Groups Along With Insulin, Compared to Insulin Alone
Description: Post-prandial blood glucose concentration in terms of mean AUC (0-120 min) was determined in subjects treated with either Exenatide 1.25 mcg or Exenatide 2.5 along with insulin, compared to insulin alone, given as a single subcutaneous injection
Time Frame: 0-120 minutes post-dose
Population: All participants who received at least one dose of each intervention and completed all study visits were included in the analyses. Only 8 subjects completed all study visits and one dropped out during the second study visit.
Measure: Mean (Standard Error); unit: mmol*L/min
Groups:
- Exenatide 1.25 mcg + Insulin: Participants who received Exenatide 1.25 mcg along with Insulin as a single subcutaneous injection
- Exenatide 2.5 mcg + Insulin: Participants who received Exenatide 2.5 mcg along with Insulin as a single subcutaneous injection
- Insulin Monotherapy: Participants who received Insulin alone as a single subcutaneous injection, part of baseline study
Arm/Group | Exenatide 1.25 mcg + Insulin | Exenatide 2.5 mcg + Insulin | Insulin Monotherapy
Number analyzed (Participants) | 8 | 8 | 8
mmol*L/min | 49 (156) | 44 (281) | 379 (259)

ADVERSE EVENTS:
Time Frame: 0-120 minutes post-dose
Groups:
- Insulin Monotherapy: Participants who received Insulin alone as a single subcutaneous injection, as part of the baseline study visit
Arm/Group | Exenatide 1.25 mcg + Insulin | Exenatide 2.5 mcg + Insulin | Insulin Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/9 | 0/9 | 0/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Exenatide 1.25 mcg + Insulin (N=9) | Exenatide 2.5 mcg + Insulin (N=9) | Insulin Monotherapy (N=9)
Hypoglycemia (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No